CLINICAL TRIAL: NCT02112734
Title: Can Vitamin D Supplementation Prevent Food Allergy in Infants? The VITALITY Trial
Brief Title: Can Vitamin D Supplementation in the First Year of Life Prevent Food Allergy in Infants? The VITALITY Trial: Parts 1&2
Acronym: VITALITY
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Murdoch Childrens Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HREC # 34168 A
Record Dates: First submitted 2014-04-10; First posted 2014-04-14 (Estimated); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Food Allergy
Keywords: vitamin D; food allergy; eczema
MeSH Terms: conditions — Food Hypersensitivity; Eczema | interventions — Vitamin D; Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- vitamin D (Active Comparator): 400 IU /daily cholecalciferol/vitamin D
  Interventions: Drug: Vitamin D
- placebo (Placebo Comparator): carrier formulation minus vitamin D
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Vitamin D — 400 IU/daily until age 12 months
  Other Names: cholecalciferol
  Arms: vitamin D
Drug: placebo — identical placebo daily
  Other Names: placebo is identical carrier minus vitamin D
  Arms: placebo

SUMMARY:
We report that Australia has the highest prevalence of Immunoglobulin(Ig)E-mediated food allergy in the world, with 10% of infants having challenge-proven food allergy in Melbourne. There has been a 5-fold increase in hospital admissions for life-threatening anaphylaxis. These changes are most pronounced in children less than 5 years, suggesting a causal role for early life determinants. We have primary data to inform hypotheses for the rise in food allergy, which appears to result from potentially modifiable factors related to the modern lifestyle, particularly Vitamin D insufficiency (VDI). We propose an intervention study to assess if infant Vitamin D supplementation during the first year of life significantly decreases the risk of early-onset food allergy and other allergic disease at 12 months (part 1) and 6 years of age (part 2). Australia is ideally placed to answer this important question since, unlike the USA, Canada and Europe, there are no population recommendations for routine infant supplementation with Vitamin D and we are one of the few developed countries that do not supplement the food chain supply with Vitamin D.

DETAILED DESCRIPTION:
There is an urgent need to prevent the onset and progression of food allergy in our population. Evidence demonstrates that food allergy and atopic eczema represent the earliest manifestations of the atopic march with 50% of infants with food allergy predicted to develop respiratory allergic diseases later in life. We report that Australia has the highest prevalence of Immunoglobulin(Ig)E-mediated food allergy in the world, with 10% of infants having challenge-proven food allergy in Melbourne. There has been a 5-fold increase in hospital admissions for life-threatening anaphylaxis. These changes are most pronounced in children less than 5 years, suggesting a causal role for early life determinants. We have primary data to inform hypotheses for the rise in food allergy, which appears to result from potentially modifiable factors related to the modern lifestyle, particularly Vitamin D insufficiency (VDI), and have demonstrated an association between VDI and increased risk of challenge-proven food allergy in 12-month old infants, which supports numerous ecological studies showing an increased risk of food allergy the further a child resides from the equator (associated with decreased UV exposure and Vitamin D levels). Despite Australia's sunny climate, population rates of VDI have steadily increased in infants and pregnant women in parallel to the apparent rise in food allergic disease. This association is biologically plausible, as there is evidence Vitamin D is critical to the healthy development of the immune system in early life. We propose an intervention study to assess if infant Vitamin D supplementation during the first year of life significantly decreases the risk of early-onset food allergy and other allergic disease at 12 months (part 1) and 6 years of age (part 2). Australia is ideally placed to answer this important question since, unlike the USA, Canada and Europe, there are no population recommendations for routine infant supplementation with Vitamin D and we are one of the few developed countries that do not supplement the food chain supply with Vitamin D.

ELIGIBILITY:
Inclusion Criteria:

Each participant must meet the following criteria to be included in this study:

* Healthy, term (born no earlier than 2 weeks before estimated date of delivery), predominantly breastfeeding infants aged 6 to 12 weeks (inclusive) who are expected to be predominantly breastfed for at least 6-months. This will be determined by answering yes/no to question 'do you intend/wish to breastfeed until your infant is at least 6 months of age.' Up to one bottle (approx. 120mL) of formula per 24 hours at the time of screening is acceptable, as this will contain <100 IU vitamin D.
* Has a parent/legally acceptable representative (LAR) capable of understanding the informed consent document and providing consent on the subject's behalf,
* The parent must expect to be able to complete 4 online questionnaires over the infant's first 12 months of life and for the infant to be available for skin prick testing (+/- food challenge) at The Royal Children's Hospital at 12 months of age.

Exclusion Criteria:

Participants meeting any of the following criteria will be excluded from the study:

* Infants who are currently receiving vitamin D supplementation
* Infants on medication that interferes with vitamin D metabolism
* Poor health due to a current or past significant disease state or congenital abnormality.
* Prematurity <37 weeks/low birth weight <2500 g/Small for gestational age (SGA)
* Unable to provide consent without the aid of an interpreter.
* Women at high risk of vitamin D deficiency with infants on vitamin D supplementation.

Ages: 6 Weeks to 12 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2739 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
The prevalence of challenge-proven food allergy at 12 months of age | At 12 months of age
  The prevalence of challenge-proven food allergy at 12 months of age determined by a positive SPT and a positive oral food challenge
The occurrence of definite food allergy or tolerance at 6 years of age | At 6 years of age
  The occurrence of definite food allergy or tolerance at 6 years of age can only be determined by combining data from an oral food challenge, a skin prick test (SPT) and/or serum specific IgE test, and/or parent/self-reported ingestion history and reactions to the index food.

SECONDARY OUTCOMES:
The prevalence of food sensitisation at 12 months of age determined by SPT positive | At 12 months of age
  The prevalence of food sensitisation at 12 months of age determined by SPT positive
The prevalence of doctor diagnosed eczema during the first postnatal year | During the first postnatal year
  The prevalence of doctor diagnosed eczema during the first postnatal year
The prevalence of vitamin D insufficiency (serum concentration of 25(OH)D <50 nmol/L ) at age 12 months determined by measuring blood taken at the 12 month clinic visit | At 12 months of age
  The prevalence of vitamin D insufficiency (serum concentration of 25(OH)D <50 nmol/L ) at age 12 months determined by measuring blood taken at the 12 month clinic visit
Allergy-related healthcare utilisation within the first 12 months of life | Within the first 12 months of life
  Allergy-related healthcare utilisation within the first 12 months of life
Infection episodes within the first 12 months of life | Within the first 12 months of life
  Infection episodes within the first 12 months of life
Measure of height at 12 months of age | At 12 months of age
  Measure of height at 12 months of age
Measure of weight at 12months of age | At 12 months of age
  Measure of weight at 12months of age
Wheeze episodes within the first 12 months of life | Within the first 12 months of life
  Wheeze episodes within the first 12 months of life
The occurrence of food sensitisation at 6 years of age determined by SPT positive | At 6 years of age
  The occurrence of food sensitisation at 6 years of age determined by SPT positive
The occurrence of asthma in the first 6 years of life | At 6 years of age
  The occurrence of asthma at 6 years of age
The occurrence of eczema in the first 6 years of life | Within first 6 years of life
  The occurrence of eczema in the first 6 years of life
The prevalence of vitamin D insufficiency (serum concentration of 25(OH)D <50 nmol/L ) at age 6 years determined by measuring blood taken at the 6 year clinic visit | At 6 years of age
  The prevalence of vitamin D insufficiency (serum concentration of 25(OH)D <50 nmol/L ) at age 6 years determined by measuring blood taken at the 6 year clinic visit
Allergy-related healthcare utilisation in the first 6 years of life | Within first 6 years of life
  Allergy-related healthcare utilisation in the first 6 years of life by data linkage from MBS and PBS
Measure of height at 6 years of age | At 6 years of age
  Measure of height at 6 years of age
Measure of Waist circumference at 6 years of age | At 6 years of age
  Measure of Waist circumference at 6 years of age
Measure of Hip circumference at 6 years of age | At 6 years of age
  Measure of Hip circumference at 6 years of age
Lung function at 6 years of age | At 6 years of age
  Lung function: bronchial responsiveness is measured using the percent change from baseline and absolute changes in forced expiratory volume (FEV) in 1 second and/or forced vital capacity (FVC) at 6 years of age
The occurrence of rhinitis in the first 6 years of life | Within first 6 years of life
  The occurrence of rhinitis in the first 6 years of life
Psychosocial Distress at 6 years of age | At 6 years of age
  Psychosocial health at 6 years of age by Kessler Psychological Distress Scale-10 (K-10) for parents The K10 scale involves 10 questions about emotional states each with a five-level response scale. Each item is scored from one 'none of the time' to five 'all of the time'. Scores of the 10 items are then summed, yielding a minimum score of 10 and a maximum score of 50. Low scores indicate low levels of psychological distress and high scores indicate high levels of psychological distress.
Psychosocial health at 6 years of age | At 6 years of age
  Psychosocial health at 6 years of age by Strengths and Difficulties Questionnaire (SDQ) for child
  SDQ ask about 25 attributes, some positive and others negative.bThese 25 items are divided between 5 scales:
  1. emotional symptoms (5 items) } 1) to 4) added together to generate a total difficulties score (based on 20 items)
  2. conduct problems (5 items)
  3. hyperactivity/inattention (5 items)
  4. peer relationship problems (5 items)
  5. prosocial behaviour (5 items)
Quality of life at 6 years of age | At 6 years of age
  Quality of life (QL) at 6 years of age by Child Health Utility 9D (CHU9D, parent proxy version; PedsQL Parent Report for Young Children ages 5-7) The questionnaire has 9 questions with 5 response levels per question. The CHU9D allows the analyst to obtain quality adjusted life years (QALYs) directly for use in cost utility analysis.
Quality of life regarding Food Allergy at 6 years of age | At 6 years of age
  Quality of life (QL) at 6 years of age by Food Allergy Quality of Life Questionnaires-Parent Form (FAQLQ-PF) All items are scored on a 7-point Likert scale from 0 (not at all troubled) to 6 (extremely troubled) [22]. The total scores are divided by the number of items answered, giving a range of scores from 0 to 6, with higher values indicating a poorer quality of life
Dental health at 6 years of age | At 6 years of age
  Dental health at 6 years of age: A registered oral health professional will examine the participant's mouth and teeth, checking for cavities/dental decay as well as developmental mark on the teeth. In addition, a 3D scan and/or photographs of the participant's teeth will be taken to document findings.

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten Perrett, MD PhD, Principal Investigator — Murdoch Childrens Research Institute
Locations (1):
- Murdoch Childrens Research Institute, Melbourne, Victoria, Australia

REFERENCES:
- [Background] Allen KJ, Koplin JJ, Ponsonby AL, Gurrin LC, Wake M, Vuillermin P, Martin P, Matheson M, Lowe A, Robinson M, Tey D, Osborne NJ, Dang T, Tina Tan HT, Thiele L, Anderson D, Czech H, Sanjeevan J, Zurzolo G, Dwyer T, Tang ML, Hill D, Dharmage SC. Vitamin D insufficiency is associated with challenge-proven food allergy in infants. J Allergy Clin Immunol. 2013 Apr;131(4):1109-16, 1116.e1-6. doi: 10.1016/j.jaci.2013.01.017. Epub 2013 Feb 27. PMID 23453797
- [Background] Allen KJ, Panjari M, Koplin JJ, Ponsonby AL, Vuillermin P, Gurrin LC, Greaves R, Carvalho N, Dalziel K, Tang ML, Lee KJ, Wake M, Curtis N, Dharmage SC. VITALITY trial: protocol for a randomised controlled trial to establish the role of postnatal vitamin D supplementation in infant immune health. BMJ Open. 2015 Dec 16;5(12):e009377. doi: 10.1136/bmjopen-2015-009377. PMID 26674499
- [Derived] Shen Z, Robert L, Stolpman M, Che Y, Allen KJ, Saffery R, Walsh A, Young A, Eckert J, Deming C, Chen Q, Conlan S, Laky K, Li JM, Chatman L, Kashaf SS; NISC Comparative Sequencing Program; VITALITY team; Kong HH, Frischmeyer-Guerrerio PA, Perrett KP, Segre JA. A genome catalog of the early-life human skin microbiome. Genome Biol. 2023 Nov 10;24(1):252. doi: 10.1186/s13059-023-03090-w. PMID 37946302